CLINICAL TRIAL: NCT06268106
Title: Graphic Novel on Anxiety and Stress in Patients Undergoing Endoscopic Ultrasound With Fine Needle Biopsy (EUS-FNB) for Pancreatic Lesions
Brief Title: Graphic Novel for Patients Undergoing EUS-FNB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB N/A
Record Dates: First submitted 2023-12-18; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anxiety; Pancreatic Cancer; Pancreatic Cystic Lesions; Stress
MeSH Terms: conditions — Anxiety Disorders; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Graphic novel will be visualized by interventional group before EUS-FNB
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard procedure informative (No Intervention): Patients in this group undergo procedure with standard explanation of the procedure itself, so they do not receive and visualize graphic novel.
- Graphic novel visualization (Experimental): Patients in this group do receive and visualize graphic novel in addition to standard explanation of the procedure.
  Interventions: Behavioral: Graphic novel visualization

INTERVENTIONS:
Behavioral: Graphic novel visualization — Patients in interventional group do receive and visualize graphic novel, which is more informative than standard informed consent.
  Arms: Graphic novel visualization

SUMMARY:
Endoscopy with endoscopic ultrasound (EUS) is a primary technique for diagnosing and treating severe pancreatic disorders. However, the procedure can cause fear and anxiety in patients, especially when a biopsy is involved. Graphic medicine, a form of visual storytelling that explores narratives of healthcare, is being used to alleviate this anxiety.

This is a prospective single-center interventional pilot study with the aim to evaluate the impact of a novel graphic on the stress and behaviors of patients with pancreatic lesions undergoing EUS-FNB. The study will run for six months with the aim to enroll patients to llok for differences in the anxiety and stress levels.

Enrolled patients will be randomly allocated to the test or control group, with the test group receiving a graphic novel to read while waiting for the procedure. Post-procedure, patients will complete the Beck Anxiety Inventory (BAI) and a modified version of the Depression Anxiety Stress Scales-21 (mDASS-21), now named mASS-14 (modified Anxiety Stress Scales-14), to assess anxiety and stress levels.

This study is conducted according to the principles of the Declaration of Helsinki regarding experimentation involving human subjects, and written informed consent will be obtained from all participants before enrollment.

DETAILED DESCRIPTION:
Endoscopy with endoscopic ultrasound (EUS) is the main technique, along with laparoscopic surgery, for diagnosing and treating severe and sometimes life-threatening pancreatic disorders. Especially in the case of pancreatic lesions, diagnostic procedures, such as EUS with fine needle biopsy (EUS-FNB), can elicit states of fear and anxiety in patients. Graphic medicine uses sequential (but not always narratively linear) visual storytelling to share health-related experiences or information.To date, there have been no applications in the field of endoscopy, so the aim of the present study is to evaluate - for the first time in the literature - the efficacy of colourful graphic novels in reducing anxiety in adult patients waiting for an endoscopic-guided biopsy for pancreatic lesions.

This is a prospective single center pilot study evaluating the impact of graphic novels on the stress and behaviour of patients with pancreatic lesions undergoing EUS-FNB at an italian tertiary referral pancreatic center. This study is being conducted according to the principles of the Declaration of Helsinki regarding experimentation involving human subjects, and written informed consent will be obtained from all participants. The authors will consecutively evaluate all patients with radiological and clinical suspicion of a pancreatic lesion from January 2024 to May 2024. After hospital admission, patients successfully enrolled and accepting participation in the study will be randomly allocated to the test or control group using dedicated software (Random Allocation Software, version 1.0) . A graphic novel will be provided to all patients in the test group, and they will be given the possibility to read it while waiting for the procedure.

The authors created a comic panel consisting of a sequence of 6 colourful vignettes in which the routine procedure of an EUS-FNB is described to the patient. The authors focused on various graphical aspects of comics, such as the facial expressions of the characters and the background, both made to look similar to the effective contexts experienced by patients at the institute. The initial drafts of the six vignettes were created using artificial intelligence and later modified by one author using graphical software.

Assessing Anxiety After EUS-FNB, all the recruited patients will receive the Beck Anxiety Inventory (BAI) and a modified version of the Depression Anxiety Stress Scales-21 (mDASS-21). Prior to the endoscopic procedures (i.e., EUS-FNB), these questionnaires will be administered anonymously in a mixed paper-pencil and/or QR Code mode to be used with a personal mobile phone. A physician, nurse or clinical assistant will be present for questions and clarification. The BAI is a 21-question self-report inventory used to assess anxiety severity in adults older than 17 years. Respondents answer questions about common anxiety symptoms, such as numbness, tingling, sweating unrelated to heat, and fear of catastrophic events. The BAI takes approximately 5 to 10 minutes to complete. Scores range from 0 (not at all) to 3 (severe), with higher scores indicating more severe anxiety. Standardized cut-offs classify anxiety levels as minimal, mild, moderate, or severe. The other questionnaire is a modified version of the DASS-21, which originally consisted of 21 items divided into three subscales (anxiety, stress and depression) with seven items each. Focusing on the anxiety and stress subscales, the questionnaire was modified in order to remove the depression subscale. Specifically, the anxiety subscale assesses physiological arousal, situational anxiety and subjective experience of the effects of anxiety, while the stress subscale evaluates chronic non-specific arousal, difficulty in relaxing, nervous tension, irritability, agitation, impatience and overactivity. Each item is rated on a 4-point scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). The total score for each subscale ranges from 0 to 14 in the modified version, with higher scores indicating higher levels of anxiety and stress. This modified version was named mDASS-21 or mASS-14. The mASS-14 has four cut-off points to classify anxiety and stress levels: normal (0-4), mild (5-8), moderate (9-11) or severe (12-14). Since the DASS-21 is a reliable and valid measure of anxiety and stress symptoms with good internal consistency, test-retest reliability and discriminant validity, this study will evaluate its modified version in this scenario. Both the BAI and mDASS-21 used in this pilot study were in the Italian versions to avoid language barriers.

Data Collection Data will be collected prospectively in a dedicated electronic case report form (eCRF) through a secure platform such as RedCap, and will include gender, age, level of education (years or diploma/degree), marital status (married/cohabiting/single), and children/grandchildren. Medical history, including previous clinically relevant conditions, such as hospitalizations, surgeries, chronic medical therapies or familiarity with cancer, will also be collected. Data regarding clinical presentation and lesion characteristics will be collected as well. The scale for intervention evaluation will be an Italian version of the Beck Anxiety Inventory (BAI), DASS-21, Cancer Worry Scale (CWS), STAI-S (State-Trait Anxiety Inventory Form) and the APAIS (Amsterdam Preoperative Anxiety and Information Scale). ECRFs in RedCap will be fully anonymized through the use of an Identification code (ID) and age instead of date of birth. ECRFs will be translated into an electronic spreadsheet for analysis.

Statistical Analysis The analysis will be performed using jamovi software (the jamovi project, version 2.3, 2023) with R language (R Core Team, 2022). Descriptive statistics will be used to analyze the patients' socio-demographic and physical characteristics. BAI and mASS-14 scores will be summarized through mean value, standard deviation (SD), maximum, median and interquartile range (IQR) as necessary. Comparisons between groups will be performed according to the most appropriate statistics (Fisher or χ-squared for categorical variables, parametric or non-parametric statistics for comparisons of continuous variables). Any relation between BAI and mASS-14 scores will be measured through a linear correlation coefficient.

ELIGIBILITY:
Inclusion criteria:

1. age ≥ 18 years
2. pancreatic solid mass or partially solid in case of cystic component
3. agree to participate in the study by signing the informed consent, and the ability to read and understand informed consent
4. patients not affected by any known psychological disorder.

Exclusion criteria:

1. patients with cognitive deficits, such that they cannot adequately complete the questionnaire and the visually impaired
2. suspected or obvious pregnancy status in female subjects
3. patients using benzodiazepines or other psychotropic medications
4. patients with previous diagnosis of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety and stress level according to BAI | up to hospital discharge, approximately up to 12 hours
  Patients will complete the Beck Anxiety Inventory (BAI) to assess anxiety and stress levels. Each variable will be scored accordingly: 0 (not at all) to 3 (severe), with higher scores indicating more severe anxiety. Standardized cut-offs classify anxiety levels as minimal (0-11), mild (12-23), moderate (24-34), or severe (35-42)
Anxiety and stress level according to mASS-14 | up to hospital discharge, approximately up to 12 hours
  Patients will complete the modified version of the Depression Anxiety Stress Scales-21 (mDASS-21), now named mASS-14, to assess anxiety and stress levels. Levels will be classified accordingly: normal (0-4), mild (5-8), moderate (9-11) or severe (12-14)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Traina, MD, Study Director — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies; Giacomo Emanuele Maria Rizzo, MD, Study Chair — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies; Ilaria Tarantino, MD, Principal Investigator — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Locations (1):
- Irccs - Ismett, Palermo, PA, Italy

IPD SHARING:
Plan to Share IPD: No